CLINICAL TRIAL: NCT03032055
Title: Validation of a Predictive Score of Acute Chest Syndrome
Acronym: Presev2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soutien aux Actions contre les Maladies du Globule Rouge (Other)
Collaborators: Theravia (Industry); Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: Presev 2 IRB 00003835
Record Dates: First submitted 2015-11-18; First posted 2017-01-26 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Vaso Occlusive Crisis; Acute Chest Syndrome
Keywords: sickle cell desease; vaso occlusive crisis; acute chest syndrome; Validation of predictif score of acute chest syndrome
MeSH Terms: conditions — Vaso-Occlusive Crises; Acute Chest Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum and DNA in Africa
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- VOC: Patients who won't develop a secondary Acute chest syndrome during a vaso occlusive crisis within 15 days after admission.
  Secondary Acute chest syndrome is defined by a new auscultatory abnormality (crepitation or bronchial breathing) OR the association of a new radiologic infiltrate and chest pain or decreased breath sounds .
  A vaso-occlusive crisis is a common painful complication of sickle cell anemia in adolescents and adults. It is a form of sickle cell crisis. Sickle cell anemia - most common in those of African, Hispanic, and Mediterranean origin - leads to sickle cell crisis when the circulation of blood vessels is obstructed by sickled red blood cells, causing ischemic injuries.
- 2°ACS: Patients who will develop a secondary acute chest syndrome during a vaso occlusive crisis within 15 days after admission.
  Secondary Acute chest syndrome is defined by a new auscultatory abnormality (crepitation or bronchial breathing) OR the association of a new radiologic infiltrate AND chest pain or decreased breath sounds .
  A vaso-occlusive crisis is a common painful complication of sickle cell anemia in adolescents and adults.It is a form of sickle cell crisis. Sickle cell anemia - most common in those of African, Hispanic, and Mediterranean origin - leads to sickle cell crisis when the circulation of blood vessels is obstructed by sickled red blood cells, causing ischemic injuries.

SUMMARY:
Vaso-Occlusive Crisis (VOC), the most common manifestation of sickle cell disease (SCD), is the first cause of death, particularly when complicated by an acute chest syndrome (ACS).

The PRESEV score could help the physicians to better manage VOC and could be used for future therapeutic trials. This predictive score of secondary ACS has to be validated in a multicenter international study.

DETAILED DESCRIPTION:
International multicentre prospective observational study.

Prediction of an ACS within 15 days after admission by the PRESEV2 score at arrival.

Validation of a Predictive Score of Acute Chest Syndrome (Presev2) associates a categorical pain score of the spine /or pelvis and 3 biological parameters: Reticulocytes, Leucocytes and Hemoglobin.

ACS is defined by crepitant or bronchial breathing or the association of new radiologic infiltrate and chest pain

Inclusion criteria:

* Children (>2 years) and adults
* Male and Female
* Homozygous SCD patients
* The patient can only be included once
* VOC admitted at the emergency unit (a severe VOC is defined as pain or tenderness affecting at least one part of the body (e.g. limbs, ribs, sternum, head (skull), spine and/or pelvis) that required hospitalization and opioids (level 3), and is not attributable to other causes.
* Patient has health care insurance (in Europe)
* Written consent given after being informed of the purpose, progress and potential risks

Exclusion criteria:

* No inaugural Acute Chest Syndrome
* Homeless patients
* Deprived of their liberty by a court or administrative order or under guardianship
* Unable to understand the purpose and conditions of carrying out the study, unable to give consent

STUDY SCHEDULE Screening and inclusion once patients are admitted at the accident and emergency department or medical day unit.

Inclusion visit (day 1) Once admitted at the accident and emergency department, the patient will be informed about the protocol and asked to participate in the study. Informed consent will be obtained according to local regulations by signing the informed consent form. The inclusion and non-inclusion criteria will be verified.

Demographic data, current and previous treatments taken within one month, and medical history will be recorded.

The following parameters of the score will be collected:

Reticulocytes and/or leucocytes counts, urea (mmol/L) and Categorical pain score.

The Score is adjusted with Hydroxyurea treatment (Yes/No) and Hb level (g/dL). Plasmodium falciparum test will be performed only in Africa. Hemoculture if fever (>38°C) is recorded within the 2 first days after admission.

Temperature, Blood pressure, Oxygen saturation, Respiratory rate, Visual analogue score will be recorded.

STUDY DURATION Inclusion period: 2 years Per patient: 15 days Total duration of the study: 2 years

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Children (>2 years) and adults
* Male and Female
* Homozygous SCD patients
* VOC admitted at the emergency unit (a severe VOC is defined as pain or tenderness affecting at least one part of the body (e.g. limbs, ribs, sternum, head (skull), spine and/or pelvis) that required hospitalization and opioids (level 3), and is not attributable to other causes.
* Patient has health care insurance (in Europe)
* Written consent given after being informed of the purpose, progress and potential risks

Exclusion criteria:

* No inaugural Acute Chest Syndrome
* Homeless patients
* Deprived of their liberty by a court or administrative order or under guardianship
* Unable to understand the purpose and conditions of carrying out the study, unable to give consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children (>2 years) and adults
  * Male and Female
  * Homozygous SCD patients
  * VOC admitted at the emergency unit (a severe VOC is defined as pain or tenderness affecting at least one part of the body (e.g. limbs, ribs, sternum, head (skull), spine and/or pelvis) that required hospitalization and opioids (level 3), and is not attributable to other causes
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure of Validation of a Predictive Score of Acute Chest Syndrome | 2 years
  The primary outcome mesure is the occurrence of an ACS defined by crepitant or bronchial breathing or the association of new radiologic infiltrats and chest pain during the first 15 days of hospitalization for Vaso Occlusive Crisis

SECONDARY OUTCOMES:
Secondary Outcome Measures: Validation of a Predictive Score of Acute Chest Syndrome | 2 years
  Association of the PRESEV 2 score with the following parameters collected for each patient:
  * The number of days of hospitalization
  * Blood transfusion requirement
  * The number of hospitalization in intensive care unit
  * Death

CONTACTS AND LOCATIONS:
Overall Officials: BARTOLUCCI Pablo, MD PhD, Pr, Principal Investigator — APHP, UPEC, INSERM
Locations (1):
- Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kassasseya C, Kene S, Besse-Hammer T, Nzouakou R, Magnang H, Telfer P, Arlet JB, de Luna G, Affo L, Dautheville S, Ngo S, Pelinski Y, Mescam C, Djoumad S, Pham Hung d'Alexandry d'Orengiani AL, Mekontso Dessap A, Michel M, Galacteros F, Audureau E, Guindo A, Habibi A, Khellaf M, Diallo D, Bartolucci P. Validation and Application of a Predictive Score of Acute Chest Syndrome. NEJM Evid. 2026 Jan;5(1):EVIDoa2500074. doi: 10.1056/EVIDoa2500074. Epub 2025 Dec 18. PMID 41410575